CLINICAL TRIAL: NCT06216028
Title: Bone Marrow Aspirate ConCentrate for the Treatment of knEe Osteoarthritis: A Phase III, muLti-centER, Pan-cAnadian, prospecTivE Trial
Brief Title: Bone Marrow Aspirate Concentrate (BMAC) Treatment for Knee Osteoarthritis
Acronym: ACCELERATE3
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CELL Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLL-001
Record Dates: First submitted 2023-12-14; First posted 2024-01-22 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Knee Osteoarthritis; Musculoskeletal Diseases
Keywords: Bone Marrow Aspirate Concentrate (BMAC); Bone Marrow Aspirate (BMA); Autologous; Phase 3; Randomized; Interventional
MeSH Terms: conditions — Osteoarthritis, Knee; Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Standard of care IA injection may include cortisone or hyaluronic acid (HA) as per discretion of the Principal Investigator
- Bone Marrow Aspirate Concentrate (BMAC) (Experimental): Cell suspension for infusion. 50 mL of Bone Marrow Aspirate collected, and 10-15 mL BMAC injected to knee(s)
  Interventions: Biological: Autologous Bone Marrow Aspirate Concentrate

INTERVENTIONS:
Biological: Autologous Bone Marrow Aspirate Concentrate — Range of between 18.7 X 104 cells/mL and 21.8 X 106 cells/mL total nucleated cells (TNC)
  Other Names: BMAC
  Arms: Bone Marrow Aspirate Concentrate (BMAC)

SUMMARY:
The purpose of the ACCELERATE3 trial is to assess the efficacy of a single intra-articular (IA) injection of autologous BMAC, in one or both knees, compared to a single IA injection of Standard of Care (SOC) in patients with mild to severe knee OA.

DETAILED DESCRIPTION:
A Pan-Canadian, Phase 3, open-label, randomized trial of bone marrow aspirate concentrate (BMAC) administration in patients with mild to severe knee OA. A total of 374 eligible patients will be randomized to BMAC or Standard of Care (SOC). Patients randomized to the interventional arm (BMAC) will have a sample of bone marrow taken (from their pelvic region) and processed at the bedside for immediate delivery back to the patient via intra-articular (IA) injection into one or both knees.

All randomized patients will be followed for 48 weeks. Blood will be collected at scheduled visits for analysis. Adverse events will be monitored throughout the trial. Assessments will be performed by physical exam and standardized questionnaires related to the physical function, health, and pain of each participant will be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥ 40 years old.
2. The subject must have a clinical diagnosis of osteoarthritis (OA) of one or both knees supported by radiological evidence (Kellgren Lawrence Grade II-IV) which is assessed locally (x-rays within the past 6 months of screening are acceptable).
3. Subjects whose knee pain persists for at least 12 weeks (about 3 months) prior to screening and does not improve symptoms with pain medications and non-operative treatment options.
4. Subject who has knee pain ≥ 40 mm out of 100 mm on single question VAS (Visual Analog Scale) at Screening (Visit 1) and prior to Randomization (Visit 2).

   Note: Subject should meet this criterion for left and right knee separately to be eligible for bilateral study treatment.
5. The subject is willing to provide written informed consent to participate in the study after reading the informed consent form and the information provided and has had the opportunity to discuss the study with the investigator or designee.
6. The subject is able to communicate satisfactorily with the investigator and to participate in, and comply with, the requirements of the study.
7. The subject is able to understand the nature of the study and any potential hazards associated with participating in it.
8. Negative pregnancy test for female subjects of childbearing potential.

Exclusion Criteria:

1. Subjects who have knee replacement surgery planned within 6 months of enrollment.
2. Subjects with a BMI ≥ 30kg/m2
3. Prior Partial Joint Replacement (PJR) or Total Joint Replacement (TJR) of one or both knees.
4. Knee surgery in the previous 6 months prior to enrollment.
5. Concomitant inflammatory disease or other condition affecting the joints (e.g., rheumatoid arthritis, septic arthritis, inflammatory joint disease, metabolic bone disease, psoriasis, gout, microcrystalline arthropathies/chondrocalcinosis, Paget's disease).
6. Congenital or acquired diseases leading to significant knee deformities that may interfere with cell application or the interpretation of results.
7. Instances of widespread pain or any pain that could interfere with the assessment of index knee pain (e.g. pain in any other part of the lower extremities, pain radiating to the knee).
8. Signs of active uncontrolled infection or known history of HIV, hepatitis, or syphilis.
9. A diagnosis of any form of cancer in the previous 6 months.
10. Actively treated with oral anticoagulants or heparin therapy (treatment such as low dose Aspirin and Plavix are allowed).
11. Participation in another clinical trial or treatment with another investigational product within 30 days prior to inclusion in the study.
12. Other conditions that may, according to medical criteria, discourage participation or impact outcome evaluation in the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
WOMAC® Pain Subscore | Change in WOMAC® Pain Subscore (Section A, Items #1-5) as measured by VAS from Baseline to the end of Week 12.
  To assess the efficacy of a single intra-articular (IA) injection of autologous BMAC, in one or both knees, compared to single IA injection of Standard of Care (SOC) in patients with mild to severe knee osteoarthritis (OA).
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). Possible score range of 0-20 for Pain (Higher scores = worse outcome).

SECONDARY OUTCOMES:
Safety (Baseline to Day 30 post IA injection) | Incidence and severity of immediate adverse events (AEs) for 30 minutes following IA injection; Incidence and severity of any AE for 30 days following IA injection; Incidence of Serious Adverse Events (SAEs)
  To assess the safety of IA injection(s) of autologous BMAC compared to SOC in patients with knee OA.
WOMAC® Physical Function Subscore | Change in WOMAC® Physical Function Subscore (Section C, Items #8-24) as measured by VAS from Baseline to the end of Week 12.
  To assess the change in the quality of life achieved by IA injection(s) of autologous BMAC compared to SOC in patients with knee OA.
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). Possible score range of 0-68 for Physical (Higher scores = worse outcome).
WOMAC® Pain Subscore | Percentage of subjects classified as 'responders' as measured by improvement in WOMAC® Pain Subscore at Week 12
  To assess the change in the quality of life achieved by IA injection(s) of autologous BMAC compared to SOC in patients with knee OA.
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). Possible score range of 0-20 for Pain (Higher scores = worse outcome).
WOMAC® Physical Function Subscore | Percentage of subjects classified as 'responders' as measured by improvement in WOMAC® Physical Function Subscore at Week 12
  To assess the change in the quality of life achieved by IA injection(s) of autologous BMAC compared to SOC in patients with knee OA.
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). Possible score range of 0-68 for Physical (Higher scores = worse outcome).
WOMAC® Physical Function and Pain Subscore | Percentage of subjects classified as 'responders' as measured by a composite responder analysis at Week 12.
  To assess the change in the quality of life achieved by IA injection(s) of autologous BMAC compared to SOC in patients with knee OA.
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). Possible score range of 0-20 for Pain and 0-68 for Physical (Higher scores = worse outcome).
WOMAC® Total Score | Change from baseline in WOMAC® Total Score (Section A, B, and C, Items #1-24) as measured by VAS at Week 12.
  To assess the change in the quality of life achieved by IA injection(s) of autologous BMAC compared to SOC in patients with knee OA.
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). Possible score range of 0-96 for a Total Score (Higher scores = worse outcome).
WOMAC® Stiffness Subscore | Change from Baseline in WOMAC® Stiffness Subscore (Section B, Items #6-7) as measured by VAS at Week 12
  To assess the change in the quality of life achieved by IA injection(s) of autologous BMAC compared to SOC in patients with knee OA.
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). Possible score range of 0-8 for Stiffness (Higher scores = worse outcome).
SF-12 | Change From Baseline in 12-Item Short-Form (SF-12) Health Survey (Quality of Life) Scores at Week 12.
  12-Item Short Form Survey (SF-12), The data calculate two summary component scores, Physical Component Summary Score (PCS) and Mental Health Component Summary Score (MCS) with eight sub-domains. Scores range from 0 to 100, where a zero score indicates the lowest level of health and 100 indicates the highest level of health, higher scores = better outcome.
  To assess the change in the quality of life achieved by IA injection(s) of autologous BMAC compared to SOC in patients with knee OA.
Six Minute Walk Test | Change from Baseline in the Six-Minute Walk Test at Week 12
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity, higher scores = better outcome To assess the change in the quality of life achieved by IA injection(s) of autologous BMAC compared to SOC in patients with knee OA.

OTHER OUTCOMES:
Exploratory - Economic | To determine the effect of IA injection(s) of autologous BMAC in promoting health economic outcomes, compared to controls
  Conduct an iterative health economic evaluation to examine the potential cost effectiveness of BMAC for the treatment of OA and the value of future research on mesenchymal stem cells (MSCs).
Exploratory - WOMAC® Pain Subscore | Change from baseline in WOMAC® Pain Subscore (Section A, Items #1-5) as measured by VAS at 24, 36, and 48-weeks
  To assess the change in the quality of life achieved by IA injection(s) of autologous BMAC compared to SOC in patients with knee OA.
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). Possible score range of 0-20 for Pain (Higher scores = worse outcome).
Exploratory - WOMAC® Physical Function Subscore | Change from baseline in WOMAC® Physical Function Subscore (Section C, Items #8-24) as measured by VAS at 24, 36, and 48-weeks
  To assess the change in the quality of life achieved by IA injection(s) of autologous BMAC compared to SOC in patients with knee OA.
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). Possible score range of 0-68 for Physical (Higher scores = worse outcome).
Exploratory - WOMAC® Total Score | Change from baseline in WOMAC® Total Score (Section A, B, and C, Items #1-24) as measured by VAS at 1, 4, 24, 36, and 48-weeks.
  To assess the change in the quality of life achieved by IA injection(s) of autologous BMAC compared to SOC in patients with knee OA.The Western Ontario and McMaster Universities Arthritis Index (WOMAC) questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). Possible score range of 0-96 for a Total Score (Higher scores = worse outcome).
Exploratory - WOMAC® Stiffness Subscore | Change from Baseline in WOMAC® Stiffness Subscore (Section B, Items #6-7) as measured by VAS at 1, 4, 24, 36, and 48-weeks.
  To assess the change in the quality of life achieved by IA injection(s) of autologous BMAC compared to SOC in patients with knee OA.
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). Possible score range of 0-8 for Stiffness (Higher scores = worse outcome).
Exploratory - SF-12 | Change From Baseline in 12-Item Short-Form (SF-12) Health Survey (Quality of Life) Scores at 4, 24, 36, and 48-weeks
  To assess the change in the quality of life achieved by IA injection(s) of autologous BMAC compared to SOC in patients with knee OA.

CONTACTS AND LOCATIONS:
Overall Officials: Riam Shamma, MD, Principal Investigator — CELL Technologies Inc.
Locations (1):
- Canadian Centres for Regenerative Therapy (CCRT), Toronto, Ontario, Canada